CLINICAL TRIAL: NCT00713635
Title: The Prenatal Effects of Congenital Heart Disease on Neurodevelopmental Outcome
Brief Title: Prenatal Effects of Congenital Heart Disease (CHD) on Neurodevelopmental Outcome
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAD1879
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Fetuses and neonates with congenital heart disease consisting of hypoplastic left heart syndrome (HLHS)
- 2: Fetuses and neonates with congenital heart disease consisting of transposition of the great arteries (TGA)
- 3: Fetuses and neonates with congenital heart disease consisting of tetralogy of fallot
- 4: Fetuses and neonates with lung masses but without congenital heart disease will serve as a control group

SUMMARY:
The purpose of this study is to investigate the prenatal impact of abnormal cardiac structure on neurodevelopmental outcomes in children with congenital heart disease.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) is the most common class of birth defect and is a major cause of infant and child death and morbidity, including neurodevelopmental delay. Children with severe forms of CHD are at high risk for a spectrum of neurocognitive difficulties that include learning disability, attention deficit and hyperactivity disorder, behavioral problems and mental retardation. The etiology of neurodevelopmental delay in children with CHD is not fully understood but is thought to be secondary to a combination of pre- and post-natal insults to the brain. It has been observed that fetuses with severe forms of CHD have abnormal blood flow to the brain as measured by Doppler ultrasound. This "centralization" or redirection of blood flow toward vital organs such as the brain has been shown to lead to abnormal brain development in other fetal diseases, such as intrauterine growth restriction. Evidence of the importance of prenatal brain development in the setting of CHD is amounting. Neonates with complex CHD demonstrate abnormalities of brain structure and blood flow prior to cardiothoracic surgery. However, to date, associations between abnormal fetal brain blood flow and neonatal neurologic outcomes and brain function have not been established in the CHD population. Finally, newborns with CHD have been shown to have abnormalities in heart rate over a 24 hour period. This finding suggests that the autonomic nervous system, which controls heart rate and blood pressure, may not function properly in infants with CHD.

The study proposes that these changes in blood flows in the fetus with heart disease could be responsible in part for poor brain growth, abnormal brain structure and function and developmental delay in childhood. Investigators will use routine obstetrical ultrasound and fetal echocardiograms to evaluate blood flow to vital organs and brain growth in fetuses with CHD. Investigators will use non-invasive fetal monitors to measure fetal heart rate and movement. Investigators will look at brain structure using Magnetic Resonance Imaging (MRI) in the fetus and newborn. Afterbirth, investigators will use non-invasive monitors to measure neonatal heart rate and blood pressure changes in response to a tilt, similar to what is experienced when placing an infant in a car seat. Investigators will use a non-invasive monitor consisting of a sticker applied to the skin to measure the level of oxygen in the brain. Investigators will also measure brain function in the newborn with an electroencephalogram(EEG) that records the electrical signaling between different parts of the brain using a special plastic hat like a swim cap. Regular physical exams with a pediatrician to measure growth and development will take place. A special test designed to detect learning disabilities will also be done when the child is 14 months old. This test will consist of talking with the child, reading stories, and showing the child pictures and colors. There will be no extra blood tests needed and none of the tests pose any risk to the mother, fetus, infant, or child.

The possible benefits to the child and the family will be early identification of any brain abnormality in the newborn period as well as learning disabilities in the toddler which will then allow the child to receive therapies designed to treat these problems. Studies show that early identification and treatment of learning disabilities are important to enhance the potential of the child.

ELIGIBILITY:
Inclusion Criteria:

1. All women who present to Columbia University Medical Center between 18-24 wks gestational age with the following fetal diagnoses will be invited to participate:
2. Hypoplastic Left Heart Syndrome (HLHS)
3. Transposition of the Great Arteries (TGA)
4. Tetralogy of Fallot (TOF)
5. Lung anomalies consisting of either congenital cystic adenomatoid malformations or bronchogenic cysts

Exclusion Criteria:

1. Documented fetal chromosomal anomaly
2. Structural brain malformations
3. Evidence of placental insufficiency or Intrauterine growth retardation
4. Documented hydrops fetalis or sustained cardiac arrhythmias
5. Anticipated delivery at an outside hospital

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study subjects will consist of mothers and infants referred to the Morgan Stanley Children's Hospital of New York-Presbyterian for evaluation of complex congenital heart disease consisting of: 1) single ventricle variant, such as hypoplastic left heart (HLHS); 2) Tetralogy of Fallot; 3) Transposition of the Great Vessels, and 4)Lung anomalies. Investigators anticipate that 24 mothers and 24 fetuses/infants will be enrolled during the period of study. This will give the study team a total of 24 women-fetus/infant dyads or 48 subjects total (if one counts the mother and the fetus/infant separately).
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2010-12; Primary Completion 2014-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental scores as measured by the Bayley Scales of Infant Development | 18 months of age

SECONDARY OUTCOMES:
Neurologic Function as defined by neonatal electroencephalographic power and coherence as measured by a neonatal high-density EEG | Neonatal EEG within 72 hours of birth
Neurologic Function as defined by fetal and neonatal autonomic nervous system assessments (fetal heart rate variability and movement coupling and neonatal tilt test) | Fetal assessment between 18-24 wk GA
Neurologic Function as defined by fetal and neonatal autonomic nervous system assessments (fetal heart rate variability and movement coupling and neonatal tilt test) | Fetal assessment between 28-32 wk GA
Neurologic Function as defined by fetal and neonatal autonomic nervous system assessments (fetal heart rate variability and movement coupling and neonatal tilt test) | Fetal assessment between 34-38 wk GA
Neurologic Function as defined by neonatal electroencephalographic power and coherence as measured by a neonatal high-density EEG | Neonatal EEG at 1 month of age

CONTACTS AND LOCATIONS:
Overall Officials: Ismee A Williams, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University College of Physicians & Surgeons, Morgan Stanley Children's Hospital of New York, New York, New York, United States